CLINICAL TRIAL: NCT04116411
Title: A Multicenter Randomized Double-blinded Controlled Phase 2 Study Evaluating the Efficacy of Valganciclovir as add-on Therapy in Glioblastoma Patients
Brief Title: A Clinical Trial Evaluating the Efficacy of Valganciclovir in Glioblastoma Patients
Acronym: VIGAS2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cecilia Soderberg-Naucler (Other)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Cecilia Soderberg-Naucler, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eudra CT: 2019-001083-30
Record Dates: First submitted 2019-08-29; First posted 2019-10-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
Keywords: cytomegalovirus; valganciclovir
MeSH Terms: conditions — Glioblastoma | interventions — Valganciclovir; Temozolomide; Radiation

STUDY DESIGN:
Intervention Model Description: A multicenter randomized double-blinded controlled phase 2 study evaluating the efficacy of valganciclovir as add-on therapy in glioblastoma patients. Patients will receive either placebo or valganciclovir according to a randomisation list, blinded to the sponsor and study team. Seven centers are aimed to include patients once approval is received for each respective study center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: VIGAS 2 is conducted under a randomised double blinded protocol. The study team and the patients are blinded to the randomisation list. Randomisation is performed by the contracted Clinical Cancer Center Unit at the Karolinska University Hospital by an unblinded person, Claudia Maes who holds responsibility to select out number codes for coded cans of the study drug. Claudia Maes is unrelated to the sponsor and the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive placebo tablets with similar appearance as the active drug. Patients receive two 450 mg tablets twice daily taken per orally for 6 weeks, thereafter two 450 mg tablet once daily for an additional 22.5 months; a total treatment time of 24 months.
  Interventions: Drug: Temozolomide 120 mg; Radiation: Radiotherapy 60 Gy; Drug: Placebo oral tablet
- Valganciclovir (Active Comparator): Patients will receive valganciclovir tablets with similar appearance as the placebo tablets. Patients receive two 450 mg valganciclovir tablets twice daily taken per orally for 6 weeks, thereafter two 450 mg valganciclovir tablets once daily for an additional 22.5 months; a total treatment time of 24 months.
  Interventions: Drug: Valganciclovir Tablets; Drug: Temozolomide 120 mg; Radiation: Radiotherapy 60 Gy

INTERVENTIONS:
Drug: Valganciclovir Tablets — Valganciclovir treatment of glioblastoma
  Other Names: Valcyte; ValGANcilovir; Valganciclovir 450 mg; J05AB14; Valganciclovir oral
  Arms: Valganciclovir
Drug: Temozolomide 120 mg — Chemotherapy
  Other Names: Temozolomide pill; Temozolomide tablet
Radiation: Radiotherapy 60 Gy — Radiation therapy
  Other Names: Radiation
Drug: Placebo oral tablet — Placebo treatment of glioblastoma
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
This study is a multicenter randomized double-blinded controlled phase 2 study evaluating the efficacy and safety of the anti-CMV drug valganciclovir vs placebo as add-on therapy in patients with glioblastoma. Valganciclovir is approved for treatment of cytomegalovirus (CMV) infections, but may also have anti-tumoral effects. Current evidence imply that most glioblastomas are CMV positive and that the virus can affect tumor aggressiveness.

DETAILED DESCRIPTION:
Adult patients will either be randomized to standard treatment (temozolomide and radiation therapy) + placebo tablets or to standard treatment + valganciclovir. Patients are randomized using 1 to 1 distribution of the patients between the treatment groups and are stratified according to methylation status of the MGMT promoter; equal proportion of patients are included in each group. A maximum of 30% of patients with methylated MGMT promoter are allowed into the study (to harmonise with current data used for statistical power calculation), as MGMT promotor methylation status is prognostic for patient survival. Patients must enter the study within 10 weeks after surgery.

Full dose treatment with 900mgs of Valganciclovir is given twice daily for 6 weeks, thereafter 900 mgs daily during 98 weeks (total treatment of 24 months). Valganciclovir is available in 450 mg tablets. The dose of Valganciclovir will be adjusted according to renal function.

This study will be performed in compliance with the protocol, ICH-GCP, the declaration of Helsinki and applicable Swedish regulatory requirements.

The study discontinuation criteria are as follows:

* Withdrawal of consent
* An adverse event which requires discontinuation of the trial medication or results in
* inability to continue to comply with trial procedures
* Disease progression which results in inability to continue to comply with trial
* procedures
* Major Protocol deviations
* Exclusion criteria met

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older
2. Patients with newly diagnosed glioblastoma, IDH 1 wt, WHO grade IV
3. Radical resection
4. Concomitant treatment with temozolomide and radiation therapy
5. MGMT promoter methylation status
6. Patients with at least KPS 70 , ECOG/WHO 2
7. Patients providing written informed consent
8. Patients cooperative and able to complete all the assessment procedures.
9. Females of child-bearing age must have a negative pregnancy test at screening (all premenopausal women, or in case when menstrual status can not be ascertained in women under the age of 55). Female patient must agree to utilize a highly efficient birth control method throughout the study period (Pearl index <1, e.g: oral contraception with gestagens, transdermal contraceptives, implants, injectables, intrauterine devices, bilateral tubal occlusion, sexual abstinence or vasectomised partner). The birth control method must be used at least 30 days after treatment end. Pregnancy testing should be performed at monthly intervals due to high teratogenic potential of valganciclovir. Men are recommended to use condoms with female partners during, and for at least 90 days following treatment with Valganciclovir.
10. Patients must be enrolled within 10 weeks after surgery

Exclusion Criteria:

1. Patients allergic to, or who do not tolerate Valganciclovir, aciclovir or valaciclovir treatment
2. Patients with decreased cognitive function (below 24 in MMSE test)
3. Pregnant or lactating females
4. Patients not signing informed consent
5. Patient is simultaneously participating in another experimental drug therapy trial
6. Neutrophil count < 1,5 cells/ 109/L
7. Platelet count < 150 cells/ 109/L
8. HGB < 80 g/L
9. Abnormal renal function (GFR < 30)
10. Secondary glioblastoma, or glioblastoma IDH1 mutated.
11. Unfit for any other reason judged by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2027-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Impact of valganciclovir on median overall survival of glioblastoma patients | Study closure at 30 months follow up. Survival analyses will be analysed at 12 and 24 months.
  Median overall survival will be analyzed using Cox regression analysis and presented by Kaplan-Meier graphs. Proportion of patients alive at 12 or 24 months, respectively, in each study arm and will be analyzed using Fisher exact test.
Baseline and demographic data | At 30 months follow up
  All baseline and demographic data will be analysed using descriptive statistics such as mean, medians, standard deviations etc. for all variables which are continuous. Variables that are categorical will be analysed using frequency tables with number of patients and percent. All these analyses will be divided by treatment group. No formal hypothesis testing will be performed for the demographic and baseline variables.

SECONDARY OUTCOMES:
Progression free survival at 12 and 24 months | 12 and 24 months
  Tumor recurrence is estimated as clinical and radiological determination (RANO criteria and NANO criteria). The progression free survival will be calculated as the (date of progression - date of first dose of study drug). Patients who are alive without progression at end of follow-up will be censored. Patients who are withdrawn from the study during the follow-up for other reason than dead will be censored at time of withdrawal. Patients who dies for any reason during the follow-up without any progression will be classified as progression using date of death as date of progression. Patients are analysed for stable disease, surgical interventions and treatment failure.
  Progression free survival will be analysed using Cox regression analysis and presented by Kaplan-Meier graphs. The difference in 12 and 24 months progression free survival rates for patients treated with valganciclovir or placebo will be analysed using Fisher exact test.
Incidence of valganciclovir treatment related adverse events | 30 months follow up time
  Number of patients with treatment related adverse events, as assessed by CTCv4. Vital signs: blood pressure (mmHg), heart rate (beats per minute), temperature (degree Celsius), clinical laboratory (total blood counts and differential analyses, liver transaminases and bilirubin, and renal function (creatinine and GFR) and physical exam. Adverse events will be analyzed using a chi-square test without continuity correction.
Health related Quality of Life using EORTC QLQ30 module | Base line and at every 3 months until 24 months follow up.
  Quality of Life measures are recoreded according to EORTC QLQ30 and BN20 module, that are validated for brain tumor patients and measured as a unit of scale. There will be a comparison of scores for patients receiving valganciclovir versus placebo treatment. These are standard tools for assessing patients reported quality of Life along time during treatment. The change from baseline will be analysed using Wilcoxon Rank Sum test.
Cognitive functions | up to 24 months
  MMSE (Mini Mental State Examination) tests are made with a questionary form and will be assesses every three months during the study. The change from baseline will be analysed using Wilcoxon Rank Sum test.
Health related Quality of Life using the EORTC BN20 module | Base line and at every 3 months until 24 months follow up.
  Quality of Life measures are recoreded according to BN20 module, that are validated for brain tumor patients and measured as a unit of scale. There will be a comparison of scores for patients receiving valganciclovir versus placebo treatment. These are standard tools for assessing patients reported quality of Life along time during treatment. The change from baseline will be analysed using Wilcoxon Rank Sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Stragliotto, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (3):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
- SE01 Karolinska University Hospital, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
When approval from authorities in Sweden allows data sharing, these will be available for other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When data is available and permissions to share these are approved, data will be available for other researchers.
Access Criteria: Access will be given by the sponsor upon request.

REFERENCES:
- [Background] Peredo I, Hellden A, Wolmer-Solberg N, Pohanka A, Stragliotto G, Rahbar A, Stahle L, Bellander BM, Soderberg-Naucler C. Ganciclovir concentrations in the cerebral extracellular space after valganciclovir treatment; a case study. BMJ Case Rep. 2015 Dec 15;2015:bcr2014207694. doi: 10.1136/bcr-2014-207694. PMID 26670887
- [Background] Rahbar A, Orrego A, Peredo I, Dzabic M, Wolmer-Solberg N, Straat K, Stragliotto G, Soderberg-Naucler C. Human cytomegalovirus infection levels in glioblastoma multiforme are of prognostic value for survival. J Clin Virol. 2013 May;57(1):36-42. doi: 10.1016/j.jcv.2012.12.018. Epub 2013 Feb 4. PMID 23391370
- [Background] Cobbs CS. Does valganciclovir have a role in glioblastoma therapy? Neuro Oncol. 2014 Mar;16(3):330-1. doi: 10.1093/neuonc/nou009. No abstract available. PMID 24523453
- [Result] Stragliotto G, Rahbar A, Solberg NW, Lilja A, Taher C, Orrego A, Bjurman B, Tammik C, Skarman P, Peredo I, Soderberg-Naucler C. Effects of valganciclovir as an add-on therapy in patients with cytomegalovirus-positive glioblastoma: a randomized, double-blind, hypothesis-generating study. Int J Cancer. 2013 Sep 1;133(5):1204-13. doi: 10.1002/ijc.28111. Epub 2013 Mar 13. PMID 23404447
- [Result] Soderberg-Naucler C, Peredo I, Stragliotto G. Valganciclovir in patients with glioblastoma. N Engl J Med. 2013 Nov 21;369(21):2066-7. doi: 10.1056/NEJMc1312413. No abstract available. PMID 24256396
- [Derived] Merchut-Maya JM, Bartek J Jr, Bartkova J, Galanos P, Pantalone MR, Lee M, Cui HL, Shilling PJ, Brochner CB, Broholm H, Maya-Mendoza A, Soderberg-Naucler C, Bartek J. Human cytomegalovirus hijacks host stress response fueling replication stress and genome instability. Cell Death Differ. 2022 Aug;29(8):1639-1653. doi: 10.1038/s41418-022-00953-w. Epub 2022 Feb 22. PMID 35194187